CLINICAL TRIAL: NCT00000320
Title: Buprenorphine Formulation Comparison: Sublingual Tablet vs. Solution
Brief Title: Buprenorphine Formulation Comparison: Sublingual Tablet vs. Solution - 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Walter Ling, M.D., Friends Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-10068-1; R01-10068-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1; liquid formulation (Active Comparator): liquid formulation
  Interventions: Drug: Buprenorphine formulation: liquid vs. tablet
- 2; tablet formulation (Active Comparator): tablet formulation
  Interventions: Drug: Buprenorphine formulation: liquid vs. tablet

INTERVENTIONS:
Drug: Buprenorphine formulation: liquid vs. tablet — random assignment to liquid buprenorphine or tablet buprenorphine
  Other Names: Subutex; Suboxone

SUMMARY:
The purpose of this study is to compare subject response to liquid vs. tablet formulations, to assess bioequivalency of liquid vs. tablet, to compare subject preference, and to evaluate if dose response curve for tablet is equal to liquid form."

DETAILED DESCRIPTION:
1) Compare subjects response to liquid vs tablet formulation 2) Assess bioequivalency of liquid vs tablet 3)Compare subject preference 4) Evaluate if dose response curve for tablet = to liquid form

ELIGIBILITY:
Inclusion Criteria:

M/F ages 18-65. Meet DMS-IV criteria for opiate dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Pregnant or nursing women. Acute medical condition that would interfere with study participation or put safety of subjects in jeopardy. Current daily use of anti-convulsants, antabuse or neuroleptics. DSM-IV diagnosis of ETOH or sedative/hypnotics dependence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 1997-10; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
blood level | across study duration

SECONDARY OUTCOMES:
drug use | across study duration
craving | across study duration
withdrawal symptoms | across study duration

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States